CLINICAL TRIAL: NCT05934357
Title: Fiber's Utilization for Energy and Life
Acronym: FUEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 24042
Record Dates: First submitted 2023-05-16; First posted 2023-07-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Diet Habit
Keywords: Fiber; Metabolizable Energy; Gastrointestinal Microbiota
MeSH Terms: conditions — Feeding Behavior | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Treatment (Experimental): Experimental treatment will contain a cereal product that contains a dietary fiber. This will be consumed three times daily for two weeks.
  Interventions: Other: Fiber
- Control treatment (Placebo Comparator): Control treatment will contain a corn meal cereal product that will be consumed three times daily for two weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Fiber — The intervention treatment will contain fiber.
  Arms: Intervention Treatment
Other: Control — The control treatment will contain corn meal.
  Arms: Control treatment

SUMMARY:
The study aims to evaluate the metabolizable energy of the typical American diet with and without the inclusion of fiber. We hypothesize that including fiber in the diet will decrease the metabolizable energy of the diet resulting in more nutrient loss into the feces and urine.

DETAILED DESCRIPTION:
The study will be a randomized, crossover, controlled feeding trial comprised of 2 experimental periods: 1) control and 2) fiber. Each experimental condition will be 16 days in length. There will be at least a 12-day compliance break between each period. Participants will undergo complete urine and fecal collection for a period five to seven days during the second half of each experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 22-75 years
* BMI between 18.5 and 39.9 kg/m2
* Ability to drop-off 1 fecal sample within 15 minutes of defecation
* Ability to pick-up meals daily
* Ability to collect fecal and urine samples daily
* Fasting glucose of <126 mg/dL

Exclusion Criteria:

* Wheat allergy or intolerance
* Any food allergies or intolerances
* Prior diagnosis of metabolic or gastrointestinal disease (kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, diabetes requiring medication)
* Women that are pregnant, had a baby within the last 12 months, or are lactating.
* Individuals that smoke, use tobacco, abuse drugs, or consume > 2 alcoholic beverages per day.
* >5% weight change in the past month or >10% change in the past year
* Oral antibiotics during the previous 6 weeks
* History of malabsorptive or restrictive bariatric surgeries (e.g., gastric bypass, sleeve gastrectomy, adjustable gastric band) or gall bladder removal surgery
* Are unable or unwilling to consume the experimental meals/snacks.
* Taking certain medications (Orlistat, bile binding resins, insulin, oral hypoglycemic agents, laxatives)
* Concurrent enrollment in another dietary, exercise, or medication study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Metabolizable Energy of the Diet | during the last 5 days of the 2 week intervention period
  The diets provided to participants will be analyzed for their energy and proximate analysis. Fecal and urine samples will be collected for 5 days during week 2 of each intervention period to calculate the total metabolizable energy of the diet. Energy and proximate analysis (dry matter, organic matter, crude protein, acid-hydrolyzed fat, and total dietary fiber) will be analyzed from the provided diet and the fecal samples. Energy will be analyzed from urine samples. The metabolizable energy content will be calculated according to the methods of Novotny et al. (2012), which considers the energy of the diet compared to the remaining energy in the collected fecal and urine samples.

SECONDARY OUTCOMES:
Fecal Microbiota | end of week 2 (end of intervention period)
  We will conduct qPCR to quantify total bacterial cells within one fresh fecal sample collected during week 2 of each condition.

OTHER OUTCOMES:
Gastrointestinal Tolerance | daily during the second week of each intervention period
  Participants will indicate if tolerance symptoms (burping, cramping/pain, distension/bloating, flatulence/gas, nausea, reflux, rumblings) are absent, mild, moderate, or severe during the second week of each intervention period. All measures will be assessed using a 4-point scale (1=absent, 2=mild, 3=moderate, 4=severe)
Bowel Function | week 2 of each intervention period
  Participants will indicate number (how many) and time of bowel movements during week 2 of each intervention condition.
Stool Consistency | daily during the second week of each intervention period
  Participants will use the Bristol Stool Scale during week 2 of each intervention condition to indicate their stool consistency.
Ease of Passage | daily during the second week of each intervention period
  Participants will indicate the ease of passage of each bowel movement during week 2 of each intervention condition. The 0-5 scale ranges from 1 (very easy) to 5 (very difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- Edward R Madigan Laboratory, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No